CLINICAL TRIAL: NCT02344238
Title: Smart Capsule for Automatic Adherence Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00030913
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Medication Adherence
Keywords: Medication compliance; Technology; Drug study
MeSH Terms: conditions — Medication Adherence | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Capsules (Other): Receive standard capsules (no ID cap technology) with compliance measured by self-report, pill count, and riboflavin measurement.
  Interventions: Dietary Supplement: Riboflavin
- ID Capsules without Prompts (Other): Receive ID capsules, with compliance measured by self-report, pill count, riboflavin measurement, and data collected by the ID Cap.
  Interventions: Other: ID Capsule; Dietary Supplement: Riboflavin
- ID Capsules with Prompts (Other): Receive ID capsules, with compliance measured by self-report, pill count, riboflavin measurement, and data collected by the ID Cap. This arm will also receive prompts (reminder calls and/or text messages) to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
  Interventions: Other: ID Capsule; Dietary Supplement: Riboflavin; Behavioral: Prompts

INTERVENTIONS:
Other: ID Capsule — Capsule containing ingestible sensor
  Arms: ID Capsules with Prompts; ID Capsules without Prompts
Dietary Supplement: Riboflavin — 50mg
Behavioral: Prompts — Reminder calls and/or text messages to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
  Arms: ID Capsules with Prompts

SUMMARY:
In pharmacotherapy trials in drug-dependent populations, medication compliance is a significant issue, as rates tend to be low and adherence to medication may predict improved outcomes (Baros et al, 2007; McRae et al, 2004; O'Brien et al, 1996; Somoza et al., 2010). However, methods commonly used to determine compliance may result in inaccurate measurement of adherence. It is therefore essential to develop measurement systems that not only accurately and objectively measure compliance, but can also have the potential to increase compliance in difficult to treat disorders such as addiction. In this study, we propose to assess the acceptability, tolerability, and efficacy of the ID-Cap System, a novel compliance measurement device, in a healthy population.

DETAILED DESCRIPTION:
The primary objective of the clinical trial is to evaluate the acceptability, tolerability, and efficacy of the ID-Cap System in a healthy population.

Participation in the study takes 10 visits over a period of approximately five weeks. The first visit is a screening visit to determine if participants are eligible to participate. After inclusion into the study, participants will be randomized into one of three groups. Participants randomized to Group 1 will have compliance measured by patient reports, pill count, and riboflavin measurement. Participants randomized to Group 2 will have compliance measured by patient reports, pill count, riboflavin measurement, and data collected by the e-Tect reader. Participants randomized to Group 3 will also have compliance measured by patient reports, pill count, riboflavin measurement, and data collected by the ID-Cap reader. However, participants randomized to this group will also receive reminder calls and/or text messages to ingest the study medication if a signal is not sent from the ID-Cap reader to the study team within one hour of the scheduled medication administration time.

After the initial screening visit, participants will present to the clinic twice weekly to complete self-reports of compliance, provide urine samples for riboflavin assessment, and be assessed for adverse effects.

They will also be asked to attend one follow-up visit to include abdominal x-ray in order to confirm passage of the capsules.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 65 years
* Must have BMI within range of 18-30
* If female and of childbearing potential, must agree to use acceptable methods of birth control for the duration of the trial
* Must consent to random assignment, and be willing to commit to medication ingestion
* Must be able to read and provide informed consent
* Must function at an intellectual level sufficient to allow accurate completion of assessments

Exclusion Criteria:

* Women who are pregnant, nursing, or plan to become pregnant during the course of the study, as abdominal X-rays will be completed on all participants
* Must not have evidence of a significant medical condition which may affect capsule passage through the gastrointestinal tract (including, but not limited to, Crohn's disease, small bowel tumors, intestinal adhesions, ulcerations, and radiation enteritis)
* Must not have past or current psychotic or bipolar disorder
* Must not be currently dependent on substances, with the exception of nicotine or caffeine, within the past 60 days
* Hypersensitivity to adhesive, riboflavin, or any capsule component
* Patients who, in the investigator's opinion, would be unable to comply with study procedures or assessments, or would be unacceptable study candidates (e.g., poses threat to staff)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, PharmD, BCPP, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Capsules: Compliance measured by self-report and riboflavin measurement.
  Riboflavin: 50mg
- ID Capsules Without Prompts: Compliance measured by self-report, riboflavin measurement, and data collected by the ID Cap.
  ID Cap: Capsule-encased computer chip
  Riboflavin: 50mg
- ID Capsules With Prompts: Compliance measured by self-report, riboflavin measurement, and data collected by the ID Cap. This arm will also receive prompts (reminder calls and/or text messages) to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
  ID Cap: Capsule-encased computer chip
  Riboflavin: 50mg
  Prompts: Reminder calls and/or text messages to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
Period: Overall Study
Arm/Group | Standard Capsules | ID Capsules Without Prompts | ID Capsules With Prompts
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Capsules | ID Capsules Without Prompts | ID Capsules With Prompts | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 9 | 34
  Male | 7 | 8 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: The primary outcome will be medication adherence as measured by percentage of doses taken among groups.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of doses taken (pill count)
Groups:
- Standard Capsules: Received standard capsules, with adherence measured by self-report, pill count and riboflavin measurement.
  Riboflavin: 50mg
- ID Capsules Without Prompts: Received ID capsules, with adherence measured by self-report, pill count, riboflavin measurement, and data collected by the ID Cap.
  ID Cap: Capsule containing ingestible sensor
  Riboflavin: 50mg
- ID Capsules With Prompts: Received ID capsules, with adherence measured by self-report, pill count, riboflavin measurement, and data collected by the ID Cap. This arm will also receive prompts (reminder calls and/or text messages) to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
  ID Cap: Capsule containing ingestible sensor
  Riboflavin: 50mg
  Prompts: Reminder calls and/or text messages to ingest the study medication if a signal is not sent to the study team within one hour of the scheduled medication administration time.
Arm/Group | Standard Capsules | ID Capsules Without Prompts | ID Capsules With Prompts
Number analyzed (Participants) | 20 | 20 | 20
percentage of doses taken (pill count) | 88.1 [82.4 to 93.7] | 96.6 [93 to 100] | 94.4 [89.5 to 99.4]

2. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: A secondary outcome will be safety and tolerability of ingestion of the ID Cap as measured by number of participants reporting adverse events in Group 1 who received standard capsules (no ID technology, study Arm 1) and Group 2 who received ID-Capsules (study Arms 2 and 3).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Standard Capsules: Received standard capsules (no ID cap technology).
- ID Capsules: Received ID capsules: capsules containing ingestible sensor
Arm/Group | Standard Capsules | ID Capsules
Number analyzed (Participants) | 20 | 40
Participants | 10 | 20

ADVERSE EVENTS:
Groups:
- Standard Capsules: Compliance measured by self-report, pill count and riboflavin measurement (study Arm 1)
  Riboflavin: 50mg
- ID Capsules: Compliance measured by self-report, pill count, riboflavin measurement, and data collected by the ID Cap (study Arms 2 and 3).
  ID Cap: Capsule-encased computer chip
  Riboflavin: 50mg
Arm/Group | Standard Capsules | ID Capsules
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/40
Other Adverse Events (participants affected / at risk) | 10/20 | 20/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Capsules (N=20) | ID Capsules (N=40)
Headache (General disorders) | 1 (2) | 2 (2)
Cold (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other GI (Gastrointestinal disorders) | 1 (1) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Allergies (General disorders) | 2 (2) | 2 (2)
Other (General disorders) | 2 (3) | 6 (7)

LIMITATIONS AND CAVEATS:
Limited generalizability- participants were primarily MUSC students & staff. The ID Cap system is only available for adherence measurement for solid oral dosage medications. Potential for user error due to the electronic nature of the ID Cap system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No